CLINICAL TRIAL: NCT06653205
Title: Systemic Inflammation Response Index and Systemic Immune Inflammation Index and Prediction of Clinical Outcome in Acute Pancreatitis
Brief Title: Prediction of Acute Pancreatitis Outcome
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Ayman Wahba, Dr, Assiut University
Other Study IDs: Acute pancreatitis outcome
Record Dates: First submitted 2024-10-20; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Acute; Pancreatitis
Keywords: Acute pancreatitis; Outcome
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of study prediction of acute pancreatitis outcome by using cheap and available laboratory resources

DETAILED DESCRIPTION:
Acute pancreatitis (AP) is a sudden inflammation of the pancreas that can vary from mild, self-resolving episodes to severe, potentially fatal conditions(1). Clinically, AP is classified into mild acute pancreatitis and severe acute pancreatitis (SAP), and SAP patients are described by multi-organ failure and high mortality rates(2). The mortality rate of acute pancreatitis varies, ranging from 3% in cases of mild edematous pancreatitis to as high as 20% in patients with pancreatic necrosis(3).The progression of AP can lead to systemic complications, making early prediction of clinical outcomes essential for effective management(4).

In recent years, there has been growing interest in identifying reliable biomarkers that can predict the severity and outcomes of acute pancreatitis(5). Systemic inflammation is a key factor in the pathophysiology of acute pancreatitis, often leading to systemic inflammatory response syndrome (SIRS) and subsequent organ dysfunction(6). Consequently, assessing systemic inflammation has become a crucial aspect of managing AP patients(7).

The Systemic Inflammation Response Index (SIRI) is recognized in the literature as an inflammatory marker that combines routine blood parameters, such as neutrophils, monocytes, and lymphocytes(8). Both SIRI and the Systemic Immune Inflammation Index (SII) are emerging as novel biomarkers for systemic inflammation(9). SIRI is calculated using neutrophil, monocyte, and lymphocyte counts, while SII is based on platelet, neutrophil, and lymphocyte counts(10)

ELIGIBILITY:
Inclusion Criteria:

Patients age >18 years old Serum amylase >3 times the upper limit of normal. abdominal pain consistent with acute pancreatitis. Typical abdominal ultrasonography and tomography findings in the routine imaging of the patients were accepted as acute pancreatitis.

Patient complaint of abdominal pain -

Exclusion Criteria:

liver diseases patients renal diseases patients malignancy patients

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient complaint of abdominal pain ,more than 18 years old,not known to have liver ,renal or malignant disease, typical abdominal ultrasound and computed tomography with findings of acute pancreatitis
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Mortality and severity of acute pancreatitis | Baseline

REFERENCES:
- [Background] Biyik M, Biyik Z, Asil M, Keskin M. Systemic Inflammation Response Index and Systemic Immune Inflammation Index Are Associated with Clinical Outcomes in Patients with Acute Pancreatitis? J Invest Surg. 2022 Aug;35(8):1613-1620. doi: 10.1080/08941939.2022.2084187. Epub 2022 Jun 5. PMID 35855674